CLINICAL TRIAL: NCT03037320
Title: Comparison of Coronally Advanced Flap and Semilunar Incision Vestibular Technique for Multiple Gingival Recessions in Maxillary Teeth - A Randomized Controlled
Brief Title: Comparison of Coronally Advanced Flap and Semilunar Incision Vestibular Technique for Multiple Gingival Recessions in Maxillary Teeth - A Randomized Controlled Trial
Acronym: CAF and SVIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indira Gandhi Institute of Dental Science (Other)
Responsible Party: Principal Investigator, Dr.Hema.P, post graduate student, Indira Gandhi Institute of Dental Science
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IGIDSIEC2016NDP28PGHPPAI
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Gingival Recession, Generalized; Root Coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): root coverage to be performed by semilunar vestibular incision technique
  Interventions: Procedure: comparison of coronally advanced flap and semilunar vestibular incision technique for root coverage in maxillary teeth
- group B (Other): root coverage by coronally advanced flap
  Interventions: Procedure: comparison of coronally advanced flap and semilunar vestibular incision technique for root coverage in maxillary teeth

INTERVENTIONS:
Procedure: comparison of coronally advanced flap and semilunar vestibular incision technique for root coverage in maxillary teeth

SUMMARY:
Comparison of Coronally advanced flap with semilunar vestibular incision technique for root coverage in patients with multiple gingival recession in maxillary teeth.

DETAILED DESCRIPTION:
the subjects attending the OPD department of periodontology, IGIDS and patients will be selected based on inclusion criteria, informed consent to be obtained from the patients,

Randomization process:

1. Patient to be selected for one of the two procedures by simple random sampling (Lottery method)
2. Baseline value will be recorded by a calibrated examiner other than the operator
3. The procedure is performed by the operator ( primary investigator)
4. Post op values to be recorded by the calibrated examiner.

Patient to be reviewed at 3 and 6 months Results will be dicussed

ELIGIBILITY:
Inclusion Criteria:

* Males and females subjects of 20-50 years.
* Patients with multiple gingival recession (2-4 teeth) of class I & II in maxillary teeth.
* Patients with well aligned teeth

Exclusion Criteria:

* Patients with class III &IV gingival recession in maxillary teeth
* Recession in relation to molars
* Patients with systemic diseases
* Medically compromised patients
* Patient with history of smoking
* Patients with erosion and root caries

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
amount of root coverage | 6 months
  root coverage in millimeters

SECONDARY OUTCOMES:
width of keratinised gingiva | 6 months
  increase of width measured in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Indira Gandhi Institute of dental sciences, Puducherry, Puducherry, India

IPD SHARING:
Plan to Share IPD: Undecided